CLINICAL TRIAL: NCT04042311
Title: High Intensity Interval Training In pATiEnts With Intermittent Claudication (INITIATE): a Proof-of-concept Prospective Cohort Study to Assess Acceptability, Feasibility and Potential Clinical Efficacy
Brief Title: High Intensity Interval Training In pATiEnts With Intermittent Claudication
Acronym: INITIATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2219
Record Dates: First submitted 2019-07-11; First posted 2019-08-01 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: Exercise; High-intensity interval training; interval training
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Workstream 1: An initial single group cohort of 30 patients will be recruited and analysed to refine/alter the intervention and exclusion criteria based on its feasibility.
  Workstream 2: This altered intervention and inclusion criteria will be considered in a further proof of concept study which will be multi-centre aiming to recruit a further x40 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Intensity interval training (workstream 1) (Experimental): High-intensity interval training performed for 20 minutes, 3 times weekly for a period of 6 weeks at 85-100% of maximal heart rate.
  Interventions: Other: High-intensity interval training

INTERVENTIONS:
Other: High-intensity interval training — a high-intensity interval training programme completed 3 times a week for 6 weeks using a stationary Wattbike.

SUMMARY:
This INITIATE study evaluates the use of high-intensity interval training as a treatment modality for patients with intermittent claudication - an ambulatory leg pain caused by narrowed arteries that supply the lower limbs.

It is an observational cohort study considering high-intensity interval training (HIIT) as a treatment for intermittent claudication, consisting of two workstreams. Workstream 1: an initial observational cohort study to consider the feasibility of the intervention and exclusion criteria. Workstream 2: a proof of concept study utilising the altered intervention and exclusion criteria following recommendations highlighted during workstream 1.

DETAILED DESCRIPTION:
Patients with peripheral vascular disease (PVD) may develop a reproducible pain in their legs when they walk, which usually subsides with rest. This is known as intermittent claudication (IC) and is caused by a reduced blood supply to the legs as a result of narrowed or hardened arteries that supply the lower limbs. This ambulatory pain impedes on activities of daily living, functional capacity and quality of life.

National Institute for Health and Care Excellence (NICE) clinical guidance recommends a 12-week supervised exercise programme as first-line treatment for IC, whereby patients are encouraged to walk to the point of maximal pain. Robust clinical trials have demonstrated that supervised exercise programmes are efficacious for improving both pain-free and maximal walking distances, whilst also potentially improving quality of life.

Despite this, supervised exercise programmes are vastly under-utilised and not always available to consultant vascular surgeons. This means that further programmes need to be developed in order to provide a range of options to patients to improve uptake and adherence rates. One such programme is a 6-week high-intensity interval training programme.

An initial observational cohort study of the 6 week HIIT programme will be conducted to determine to determine the feasibility of the intervention and inclusion criteria. The results from this will be used to make any necessary changes to the HIIT intervention before moving into a proof of concept study, considering the utility, safety, acceptability and potential clinical efficacy of this programme.

ELIGIBILITY:
Workstream 1

Inclusion criteria:

* Aged >18 years
* Ankle-brachial pressure index (ABPI) <0.9 at rest or a systolic pressure drop of ≥20mmHg at the ankle after exercise testing
* Ability to walk unaided
* English speaking and able to comply with exercise instructions

Exclusion criteria:

* Unable to provide informed consent
* Critical limb threatening ischaemia / rest pain / tissue loss
* Active cancer treatment
* Significant comorbidities precluding safe participation in exercise testing and / or training according to the American College of Sports Medicine (ACSM) guidelines (28)
* Resting/uncontrolled tachycardia (>100 beats per minute [bpm]) and/or resting/uncontrolled hypertension (systolic blood pressure >180 millimetres of mercury [mmHg] or diastolic blood pressure >100mmHg)
* Symptomatic hypotension

Additional exclusion criteria:

Following baseline cardiopulmonary exercise test (CPET), patients will be withdrawn and prevented from continuing their involvement in the study if there is any evidence of:

* Exercise-induced myocardial ischaemia or significant haemodynamic compromise (manifesting as anginal symptoms, significant ECG changes or an abnormal blood pressure response).
* An inability to complete a maximal effort CPET

Workstream 2:

Inclusion criteria:

* Aged >18 years
* ABPI <0.9 at rest or a systolic pressure drop of ≥20mmHg at the ankle after exercise testing
* Ability to walk unaided
* English speaking and able to comply with exercise instructions

Exclusion criteria:

* Unable to provide informed consent
* Critical limb threatening ischaemia / rest pain / tissue loss
* Active cancer treatment
* Significant comorbidities precluding safe participation in exercise testing and / or training according to the American College of Sports Medicine (ACSM) guidelines (28)
* Resting/uncontrolled tachycardia (>100bpm) and/or resting/uncontrolled hypertension (systolic blood pressure >180mmHg or diastolic blood pressure >100mmHg)
* Symptomatic hypotension

Additional exclusion criteria:

Following baseline CPET, patients will be withdrawn and prevented from continuing their involvement in the study if there is any evidence of:

● Exercise-induced myocardial ischaemia or significant haemodynamic compromise (manifesting as anginal symptoms, significant ECG changes or an abnormal blood pressure response).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Pymer, MSc, Principal Investigator — Academic Vascular Surgical Unit, Hull York Medical School
Locations (1):
- Academic Vascular Surgical Unit, Vascular Dept. 1st Floor Tower Block, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pymer S, Harwood AE, Ibeggazene S, McGregor G, Huang C, Nicholls AR, Ingle L, Long J, Rooms M, Chetter IC, Twiddy M. High INtensity Interval Training in pATiEnts with Intermittent Claudication: A Qualitative Acceptability Study. Ann Vasc Surg. 2024 May;102:17-24. doi: 10.1016/j.avsg.2023.11.043. Epub 2024 Jan 30. PMID 38301846
- [Result] Pymer S, Harwood AE, Prosser J, Waddell A, Rhavindhran B, Ibeggazene S, McGregor G, Huang C, Twiddy M, Nicholls AR, Ingle L, Carroll S, He H, Long J, Rooms M, Chetter IC. High-intensity interval training in patients with intermittent claudication. J Vasc Surg. 2023 Oct;78(4):1048-1056.e4. doi: 10.1016/j.jvs.2023.05.045. Epub 2023 Jun 16. PMID 37330704
- [Derived] Pymer S, Ibeggazene S, Palmer J, Smith GE, Harwood AE, Carroll S, Ingle L, Chetter IC. Considering the Feasibility, Tolerability, and Safety of High-Intensity Interval Training as a Novel Treatment for Patients With Intermittent Claudication. J Cardiopulm Rehabil Prev. 2021 May 1;41(3):188-193. doi: 10.1097/HCR.0000000000000551. PMID 33186201
- [Derived] Pymer S, Harwood A, Ibeggazene S, McGregor G, Huang C, Twiddy M, Nicholls AR, Ingle L, Carroll S, Long J, Rooms M, Chetter IC; INITIATE investigator group. High INtensity Interval Training In pATiEnts with intermittent claudication (INITIATE): protocol for a multicentre, proof-of-concept, prospective interventional study. BMJ Open. 2020 Jul 6;10(7):e038825. doi: 10.1136/bmjopen-2020-038825. PMID 32636290

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Intensity Interval Training: High-intensity interval training performed for 20 minutes, 3 times weekly for a period of 6 weeks at 85-100% of maximal heart rate.
Period: Overall Study
Arm/Group | High-Intensity Interval Training
Started | 70
Participants Enrolled in Workstream 1 | 30
Participants Completing Workstream 1 | 15
Participants Enrolled in Workstream 2 | 40
Participants Completing Workstream 2 | 31
Completed | 46
Not Completed | 24
Not completed — Abnormal cardiopulmonary exercise test (CPET) or unable to achieve a maximal test | 9
Not completed — Unable to tolerate | 4
Not completed — Concurrent illness | 2
Not completed — Adverse Event | 2
Not completed — No longer meeting inclusion criteria | 2
Not completed — No reason given | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics broken down by workstream
Groups:
- High-Intensity Interval Training (Workstream 2): High-intensity interval training performed for 20 minutes, 3 times weekly for a period of 6 weeks at 85-100% of maximal heart rate
- Total: Total of all reporting groups
Arm/Group | High-Intensity Interval Training (Workstream 1) | High-Intensity Interval Training (Workstream 2) | Total
Number analyzed (Participants) | 30 | 40 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] — Workstream 1, n=30 Workstream 2, n=40 Population: Workstream 1, n=30 Workstream 2, n=40
  years | 69 (9) | 69 (8) | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Workstream 1, n=30 Workstream 2, n=40
  Participants
    Female | 7 | 5 | 12
    Male | 23 | 35 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] — Population: Workstream 1, n=30 Workstream 2, n=40
  cm | 168.5 (7.2) | 169.1 (10.0) | 168.7 (8.3)
Weight [Mean (Standard Deviation); unit: kg] — Population: Workstream 1, n=30 Workstream 2, n=40
  kg | 81.6 (16.2) | 79.9 (14.5) | 80.6 (15.2)
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Workstream 1, n=30 Workstream 2, n=40
  kg/m^2 | 28.5 (4.0) | 28.0 (3.9) | 28.2 (3.9)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Workstream 1, n=30 Workstream 2, n=40
  mmHg | 146 (20) | 146 (20) | 146 (19)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Workstream 1, n=30 Workstream 2, n=40
  mmHg | 79 (8) | 81 (13) | 80 (11)
Ankle-brachial pressure index (ABPI) (worst leg) [Mean (Standard Deviation); unit: Index] — ABPI involves measuring the systolic blood pressure in the brachial, dorsalis pedis and posterial tibial arteries bilaterally using an appropriately sized sphygmomanometer, placed on the arms and above the ankles. The ABPI is calculated by dividing the highest systolic pressure of the dorsalis pedis and posterior tibial arteries of each ankle by the highest systolic brachial pressure of both arms. Population: Workstream 1, n=30 Workstream 2, n=40
  Index | 0.64 (0.20) | 0.63 (0.21) | 0.63 (.21)
Intermittent claudication distance (ICD) [Mean (Standard Deviation); unit: metres] — Population: Workstream 1, n=30 Workstream 2, n=40
  metres | 118.6 (109.9) | 130.2 (88.8) | 125.1 (97.9)
Maximum Walking Distance (MWD) [Mean (Standard Deviation); unit: metres] — Population: Workstream 1, n=30 Workstream 2, n=40
  metres | 283 (190.5) | 327.5 (206.8) | 307.9 (199.6)
Smoking status [Count of Participants; unit: Participants] — Population: Workstream 1, n=30 Workstream 2, n=40
  Participants
    Current | 11 | 13 | 24
    Ex | 17 | 22 | 39
    Non-smoker | 2 | 5 | 7
Best medical therapy (BMT) [Count of Participants; unit: Participants] — Best medical therapy comprised being prescribed an antiplatelet or anticoagulant and a statin. Population: Workstream 1, n=30 Workstream 2, n=40
  Participants | 26 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Test - Related Withdrawals
Description: Defined by examining the number of withdrawals related to the intervention or study procedures (i.e. patients unable to tolerate).
Time Frame: From the first to last exercise session, i.e. from week 0 to week 6.
Population: Workstream 1 = 30 participants Workstream 2 = 40 participants
Measure: Count of Participants; unit: Participants
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 70
Participants
  Workstream 1 - unable to tolerate HIIT or CPEX: number analyzed (Participants) | 30
  Workstream 1 - unable to tolerate HIIT or CPEX | 1
  Workstream 2 - unable to tolerate HIIT or CPEX: number analyzed (Participants) | 40
  Workstream 2 - unable to tolerate HIIT or CPEX | 3

2. Primary Outcome: Feasibility Test
Description: Feasibility measures included the number of patients screened vs. the number eligible, the number of patients eligible vs. the number recruited and the number recruited vs. the number completed.
Time Frame: From study opening to completion/withdrawal of the last patient
Population: The overall number of participants analysed in the number of patients screened. Each row then represents the number of patients eligible vs. screened, the number recruited vs. eligible and the number completed vs. recruited.
Measure: Number; unit: participants
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 424
participants
  Workstream 1 - screened: number analyzed (Participants) | 144
  Workstream 1 - screened | 144
  Workstream 1 - eligible: number analyzed (Participants) | 144
  Workstream 1 - eligible | 95
  Workstream 1 - recruited: number analyzed (Participants) | 95
  Workstream 1 - recruited | 30
  Workstream 1 - completed: number analyzed (Participants) | 30
  Workstream 1 - completed | 15
  Workstream 2 - screened: number analyzed (Participants) | 280
  Workstream 2 - screened | 280
  Workstream 2 - eligible: number analyzed (Participants) | 280
  Workstream 2 - eligible | 165
  Workstream 2 - recruited: number analyzed (Participants) | 165
  Workstream 2 - recruited | 40
  Workstream 2 - completed: number analyzed (Participants) | 40
  Workstream 2 - completed | 31

3. Primary Outcome: Tolerability Test - Achieving the Required Intensity
Description: Considers the patients ability to achieve and maintain exercise at the appropriate intensity for the duration of each session
Time Frame: From the first to last exercise session, i.e. from week 0 to week 6.
Population: Includes all participants that completed the programme and the type of units is the number of HIIT intervals completed. The number analysed is the total amount of intervals completed per workstream. The count of units is the number of intervals where the required intensity was achieved.
Measure: Count of Units; unit: Number of HIIT intervals
Units Other Than Participants: Number of HIIT intervals
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 46
Number analyzed (Number of HIIT intervals) | 7998
Number of HIIT intervals
  Workstream 1 - intervals at the required intensity: number analyzed (Participants) | 15
  Workstream 1 - intervals at the required intensity: number analyzed (Number of HIIT intervals) | 2576
  Workstream 1 - intervals at the required intensity | 2210
  Workstream 2 - intervals at the required intensity: number analyzed (Participants) | 31
  Workstream 2 - intervals at the required intensity: number analyzed (Number of HIIT intervals) | 5422
  Workstream 2 - intervals at the required intensity | 4546

4. Primary Outcome: Tolerability Test - Number of Sessions Completed
Description: Considers the number of sessions completed compared to the theoretical number.
Time Frame: From the first to last exercise session, i.e. from week 0 to week 6.
Population: Includes all participants that completed the programme and the type of units is the number of HIIT sessions completed. The number analysed is the total amount of planned sessions per workstream. The count of units is the number of sessions that were actually attended.
Measure: Count of Units; unit: Number of HIIT sessions
Units Other Than Participants: Number of HIIT sessions
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 46
Number analyzed (Number of HIIT sessions) | 828
Number of HIIT sessions
  Workstream 1 - HIIT sessions completed: number analyzed (Participants) | 15
  Workstream 1 - HIIT sessions completed: number analyzed (Number of HIIT sessions) | 270
  Workstream 1 - HIIT sessions completed | 270
  Workstream 2 - HIIT sessions completed: number analyzed (Participants) | 31
  Workstream 2 - HIIT sessions completed: number analyzed (Number of HIIT sessions) | 558
  Workstream 2 - HIIT sessions completed | 551

5. Primary Outcome: Tolerability Test - Number of HIIT Intervals Completed
Description: Considers the number of HIIT intervals completed compared to the theoretical number.
Time Frame: From the first to last exercise session, i.e. from week 0 to week 6.
Population: Includes all participants that completed the programme and the type of units is the number of HIIT intervals completed. The number analysed is the total amount of planned HIIT intervals. The count of units is the number of intervals that were actually completed.
Measure: Count of Units; unit: Number of HIIT intervals
Units Other Than Participants: Number of HIIT intervals
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 46
Number analyzed (Number of HIIT intervals) | 828
Number of HIIT intervals
  Workstream 1 - HIIT intervals completed: number analyzed (Participants) | 15
  Workstream 1 - HIIT intervals completed: number analyzed (Number of HIIT intervals) | 270
  Workstream 1 - HIIT intervals completed | 234
  Workstream 2 - HIIT intervals completed: number analyzed (Participants) | 31
  Workstream 2 - HIIT intervals completed: number analyzed (Number of HIIT intervals) | 558
  Workstream 2 - HIIT intervals completed | 475

6. Secondary Outcome: Safety Events Recorded
Description: Defined as the occurrence of any adverse or serious adverse events related to the intervention.
Time Frame: From enrolment to completion of 12-week follow-up
Population: The analysed population is all patients who were recruited to the programme. Adverse events were considered at each visit and exercise session.
Measure: Number; unit: Events
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 70
Events
  Workstream 1: number analyzed (Participants) | 30
  Workstream 1 | 3
  Workstream 2: number analyzed (Participants) | 40
  Workstream 2 | 9

7. Secondary Outcome: Acceptability Testing
Description: An evaluation of the acceptability of the exercise intervention assessed by patient feedback, using semi-structured interviews.
Time Frame: post-intervention follow-up, i.e. week 6.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 23
Participants | 23

8. Secondary Outcome: Maximum Walking Distance
Description: assessment of the distance that the patient can currently walk before having to stop due to claudication pain.
Time Frame: Baseline, post-intervention (week 6), then 4 weeks (week 10) and 12 weeks (week 18) post-intervention.
Population: Only patients completing the programme and providing baseline and follow-up data are included. This comprises:
  Post-intervention follow-up Workstream 1; n = 15/30 Workstream 2; n = 29/40 Total = 44/70.
  4-week post-intervention follow-up Workstream 1; n = 12/30 Workstream 2; n = 16/40 Total = 28/70.
  12-week post-intervention follow-up Workstream 1; n =11/30 Workstream 2; n = 24/40 Total = 35/70.
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 44
metres
  Workstream 1 baseline: number analyzed (Participants) | 15
  Workstream 1 baseline | 243.8 (102.2)
  Workstream 1 Post-intervention follow-up: number analyzed (Participants) | 15
  Workstream 1 Post-intervention follow-up | 365.2 (153.6)
  Workstream 1 - 4-week post intervention follow-up: number analyzed (Participants) | 12
  Workstream 1 - 4-week post intervention follow-up | 365.4 (172.3)
  Workstream 1 - 12-week post intervention follow-up: number analyzed (Participants) | 11
  Workstream 1 - 12-week post intervention follow-up | 374.2 (233.4)
  Workstream 2 baseline: number analyzed (Participants) | 29
  Workstream 2 baseline | 366.5 (201.0)
  Workstream 2 Post-intervention follow-up: number analyzed (Participants) | 29
  Workstream 2 Post-intervention follow-up | 455.0 (220.8)
  Workstream 2 - 4-week post intervention follow-up: number analyzed (Participants) | 16
  Workstream 2 - 4-week post intervention follow-up | 450.7 (242.8)
  Workstream 2 - 12-week post intervention follow-up: number analyzed (Participants) | 24
  Workstream 2 - 12-week post intervention follow-up | 448.1 (240.9)

9. Secondary Outcome: Peak Oxygen Uptake
Description: Peak oxygen uptake assessed via cardiopulmonary exercise testing
Time Frame: Baseline, post-intervention (week 6), then 4 weeks (week 10) and 12 weeks (week 18) post-intervention.
Population: Only patients completing the programme and providing baseline and follow-up data are included. This comprises:
  End of programme follow-up:
  Workstream 1; n = 13/30 Workstream 2; n = 29/40 Total = 42/70.
  4-week follow-up: Workstream 1; n = 10/30 Workstream 2; n = 16/40 Total = 26/70.
  12-week follow-up: Workstream 1; n = 9/30 Workstream 2; n = 20/40 Total = 29/70.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 42
ml/kg/min
  Workstream 1 - baseline VO2Peak: number analyzed (Participants) | 13
  Workstream 1 - baseline VO2Peak | 15.4 (2.8)
  Workstream 1 - post-intervention follow-up VO2Peak: number analyzed (Participants) | 13
  Workstream 1 - post-intervention follow-up VO2Peak | 15.9 (3.0)
  Workstream 1 - 4-week post-intervention follow-up VO2Peak: number analyzed (Participants) | 10
  Workstream 1 - 4-week post-intervention follow-up VO2Peak | 15.8 (2.3)
  Workstream 1 - 12-week post-intervention follow-up VO2Peak: number analyzed (Participants) | 9
  Workstream 1 - 12-week post-intervention follow-up VO2Peak | 15.3 (3.1)
  Workstream 2 - baseline VO2Peak: number analyzed (Participants) | 29
  Workstream 2 - baseline VO2Peak | 16.4 (3.9)
  Workstream 2 - post-intervention follow-up VO2Peak: number analyzed (Participants) | 29
  Workstream 2 - post-intervention follow-up VO2Peak | 17.1 (4.3)
  Workstream 2 - 4-week post-intervention follow-up VO2Peak: number analyzed (Participants) | 16
  Workstream 2 - 4-week post-intervention follow-up VO2Peak | 16.9 (4.6)
  Workstream 2 - 12-week post-intervention follow-up VO2Peak: number analyzed (Participants) | 20
  Workstream 2 - 12-week post-intervention follow-up VO2Peak | 17.8 (4.1)

10. Secondary Outcome: Quality of Life Questionnaire Short-form-36 (SF-36)
Description: Patient reported quality of life using the SF-36 SF-36 is a 36-Item Short Form Health Survey questionnaire. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Time Frame: Baseline and post-intervention (week 6)
Population: Only patients completing the programme and providing baseline and follow-up data are included. This comprises:
  Workstream 1; n = 15/30 Workstream 2; n = 30/40 Total = 45/70.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 45
units on a scale
  Workstream 1 baseline physical functioning: number analyzed (Participants) | 15
  Workstream 1 baseline physical functioning | 50.1 (18.2)
  Workstream 1 follow-up physical functioning: number analyzed (Participants) | 15
  Workstream 1 follow-up physical functioning | 54.7 (20.2)
  Workstream 1 baseline role physical: number analyzed (Participants) | 15
  Workstream 1 baseline role physical | 52.5 (26.9)
  Workstream 1 follow-up role physical: number analyzed (Participants) | 15
  Workstream 1 follow-up role physical | 55.4 (27.7)
  Workstream 1 baseline pain: number analyzed (Participants) | 15
  Workstream 1 baseline pain | 47.9 (13.9)
  Workstream 1 follow-up pain: number analyzed (Participants) | 15
  Workstream 1 follow-up pain | 50.0 (22.6)
  Workstream 1 baseline general health: number analyzed (Participants) | 15
  Workstream 1 baseline general health | 46.6 (19.9)
  Workstream 1 follow-up general health: number analyzed (Participants) | 15
  Workstream 1 follow-up general health | 52.7 (20.8)
  Workstream 1 baseline vitality: number analyzed (Participants) | 15
  Workstream 1 baseline vitality | 41.5 (15.2)
  Workstream 1 follow-up vitality: number analyzed (Participants) | 15
  Workstream 1 follow-up vitality | 50.9 (17.4)
  Workstream 1 baseline social functioning: number analyzed (Participants) | 15
  Workstream 1 baseline social functioning | 76.8 (26.3)
  Workstream 1 follow-up social functioning: number analyzed (Participants) | 15
  Workstream 1 follow-up social functioning | 76.8 (27.2)
  Workstream 1 baseline role emotional: number analyzed (Participants) | 15
  Workstream 1 baseline role emotional | 73.3 (30.2)
  Workstream 1 follow-up role emotional: number analyzed (Participants) | 15
  Workstream 1 follow-up role emotional | 80.0 (25.2)
  Workstream 1 baseline mental health: number analyzed (Participants) | 15
  Workstream 1 baseline mental health | 68.6 (17.7)
  Workstream 1 follow-up mental health: number analyzed (Participants) | 15
  Workstream 1 follow-up mental health | 73.6 (17.8)
  Workstream 1 baseline PCS: number analyzed (Participants) | 15
  Workstream 1 baseline PCS | 37.8 (7.6)
  Workstream 1 follow-up PCS: number analyzed (Participants) | 15
  Workstream 1 follow-up PCS | 39.4 (7.3)
  Workstream 1 baseline MCS: number analyzed (Participants) | 15
  Workstream 1 baseline MCS | 49.2 (9.9)
  Workstream 1 follow-up MCS: number analyzed (Participants) | 15
  Workstream 1 follow-up MCS | 51.9 (9.4)
  Workstream 2 baseline physical functioning: number analyzed (Participants) | 30
  Workstream 2 baseline physical functioning | 53.3 (19.2)
  Workstream 2 follow-up physical functioning: number analyzed (Participants) | 30
  Workstream 2 follow-up physical functioning | 56.2 (19.1)
  Workstream 2 baseline role physical: number analyzed (Participants) | 30
  Workstream 2 baseline role physical | 52.9 (23.9)
  Workstream 2 follow-up role physical: number analyzed (Participants) | 30
  Workstream 2 follow-up role physical | 60.8 (24.7)
  Workstream 2 baseline pain: number analyzed (Participants) | 30
  Workstream 2 baseline pain | 47.3 (19.9)
  Workstream 2 follow-up pain: number analyzed (Participants) | 30
  Workstream 2 follow-up pain | 54.1 (22.6)
  Workstream 2 baseline general health: number analyzed (Participants) | 30
  Workstream 2 baseline general health | 54.4 (21.2)
  Workstream 2 follow-up general health: number analyzed (Participants) | 30
  Workstream 2 follow-up general health | 54.8 (19.3)
  Workstream 2 baseline vitality: number analyzed (Participants) | 30
  Workstream 2 baseline vitality | 53.2 (17.8)
  Workstream 2 follow-up vitality: number analyzed (Participants) | 30
  Workstream 2 follow-up vitality | 55.8 (19.3)
  Workstream 2 baseline social functioning: number analyzed (Participants) | 30
  Workstream 2 baseline social functioning | 77.5 (24.7)
  Workstream 2 follow-up social functioning: number analyzed (Participants) | 30
  Workstream 2 follow-up social functioning | 75.4 (27.9)
  Workstream 2 baseline role emotional: number analyzed (Participants) | 30
  Workstream 2 baseline role emotional | 73.1 (25.2)
  Workstream 2 follow-up role emotional: number analyzed (Participants) | 30
  Workstream 2 follow-up role emotional | 75.6 (25.3)
  Workstream 2 baseline mental health: number analyzed (Participants) | 30
  Workstream 2 baseline mental health | 76.7 (14.5)
  Workstream 2 follow-up mental health: number analyzed (Participants) | 30
  Workstream 2 follow-up mental health | 76.7 (19.8)
  Workstream 2 baseline PCS: number analyzed (Participants) | 30
  Workstream 2 baseline PCS | 38.5 (7.0)
  Workstream 2 follow-up PCS: number analyzed (Participants) | 30
  Workstream 2 follow-up PCS | 40.7 (7.3)
  Workstream 2 baseline MCS: number analyzed (Participants) | 30
  Workstream 2 baseline MCS | 52.3 (8.8)
  Workstream 2 follow-up MCS: number analyzed (Participants) | 30
  Workstream 2 follow-up MCS | 52 (10.4)

11. Secondary Outcome: Vascular Quality of Life Questionnaire - (VascuQol)
Description: VascuQoL includes 25 items subdivided into 5 domains and a sum score is also calculated by dividing the total score by 25.
  Each domain and the total score range from 1 to 7 with 1 representing the worst score and 7 the best.
Time Frame: Baseline and post-intervention (week 6) follow-up
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 45
units on a scale
  Workstream 1 baseline pain score: number analyzed (Participants) | 15
  Workstream 1 baseline pain score | 4.2 (1.3)
  Workstream 1 follow-up pain score: number analyzed (Participants) | 15
  Workstream 1 follow-up pain score | 4.4 (1.5)
  Workstream 1 baseline social score: number analyzed (Participants) | 15
  Workstream 1 baseline social score | 5.5 (1.7)
  Workstream 1 follow-up social score: number analyzed (Participants) | 15
  Workstream 1 follow-up social score | 5.7 (1.0)
  Workstream 1 baseline activities score: number analyzed (Participants) | 15
  Workstream 1 baseline activities score | 4.4 (1.2)
  Workstream 1 follow-up activities score: number analyzed (Participants) | 15
  Workstream 1 follow-up activities score | 4.6 (1.0)
  Workstream 1 baseline symptom score: number analyzed (Participants) | 15
  Workstream 1 baseline symptom score | 5.5 (0.6)
  Workstream 1 follow-up symptom score: number analyzed (Participants) | 15
  Workstream 1 follow-up symptom score | 5.8 (0.6)
  Workstream 1 baseline emotional score: number analyzed (Participants) | 15
  Workstream 1 baseline emotional score | 5.4 (1.6)
  Workstream 1 follow-up emotional score: number analyzed (Participants) | 15
  Workstream 1 follow-up emotional score | 5.4 (1.4)
  Workstream 1 baseline total score: number analyzed (Participants) | 15
  Workstream 1 baseline total score | 4.9 (1.1)
  Workstream 1 follow-up total score: number analyzed (Participants) | 15
  Workstream 1 follow-up total score | 5.1 (1.0)
  Workstream 2 baseline pain score: number analyzed (Participants) | 30
  Workstream 2 baseline pain score | 3.7 (1.2)
  Workstream 2 follow-up pain score: number analyzed (Participants) | 30
  Workstream 2 follow-up pain score | 4.5 (1.1)
  Workstream 2 baseline social score: number analyzed (Participants) | 30
  Workstream 2 baseline social score | 5.2 (1.7)
  Workstream 2 follow-up social score: number analyzed (Participants) | 30
  Workstream 2 follow-up social score | 5.4 (1.8)
  Workstream 2 baseline activities score: number analyzed (Participants) | 30
  Workstream 2 baseline activities score | 4.3 (1.2)
  Workstream 2 follow-up activities score: number analyzed (Participants) | 30
  Workstream 2 follow-up activities score | 4.7 (1.2)
  Workstream 2 baseline symptom score: number analyzed (Participants) | 30
  Workstream 2 baseline symptom score | 4.9 (1.3)
  Workstream 2 follow-up symptom score: number analyzed (Participants) | 30
  Workstream 2 follow-up symptom score | 5.4 (1.0)
  Workstream 2 baseline emotional score: number analyzed (Participants) | 30
  Workstream 2 baseline emotional score | 5.2 (1.3)
  Workstream 2 follow-up emotional score: number analyzed (Participants) | 30
  Workstream 2 follow-up emotional score | 5.5 (1.4)
  Workstream 2 baseline total score: number analyzed (Participants) | 30
  Workstream 2 baseline total score | 4.6 (1.1)
  Workstream 2 follow-up total score: number analyzed (Participants) | 30
  Workstream 2 follow-up total score | 5.0 (1.1)

12. Secondary Outcome: Ankle-Brachial Pressure Index
Description: The index or ratio of the pressure in the ankle compared with the arm.
Time Frame: Baseline, post-intervention (week 6), then 4 weeks (week 10) and 12 weeks (week 18) post-intervention.
Population: Only patients completing the programme and providing baseline and follow-up data are included. This comprises:
  Post-intervention follow-up Workstream 1; n = 15/30 Workstream 2; n = 30/40 Total = 44/70.
  4-week post-intervention follow-up Workstream 1; n = 12/30 Workstream 2; n = 16/40 Total = 28/70.
  12-week post-intervention follow-up Workstream 1; n =11/30 Workstream 2; n = 24/40 Total = 35/70.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 45
Index
  Workstream 1 baseline: number analyzed (Participants) | 15
  Workstream 1 baseline | 0.76 (0.22)
  Workstream 1 post- intervention follow-up: number analyzed (Participants) | 15
  Workstream 1 post- intervention follow-up | 0.78 (0.19)
  Workstream 1 - 4-week post-intervention follow-up: number analyzed (Participants) | 12
  Workstream 1 - 4-week post-intervention follow-up | 0.74 (0.20)
  Workstream 1 - 12-week post-intervention follow-up: number analyzed (Participants) | 11
  Workstream 1 - 12-week post-intervention follow-up | 0.80 (0.20)
  Workstream 2 baseline: number analyzed (Participants) | 30
  Workstream 2 baseline | 0.74 (0.19)
  Workstream 2 post-intervention follow-up: number analyzed (Participants) | 30
  Workstream 2 post-intervention follow-up | 0.76 (0.14)
  Workstream 2 - 4-week post-intervention follow-up: number analyzed (Participants) | 16
  Workstream 2 - 4-week post-intervention follow-up | 0.78 (0.12)
  Workstream 2 - 12-week post-intervention follow-up: number analyzed (Participants) | 24
  Workstream 2 - 12-week post-intervention follow-up | 0.74 (0.14)

13. Secondary Outcome: Peak Power Output
Description: Peak power output assessed via CPET
Time Frame: Baseline, post-intervention (week 6), then 4 weeks (week 10) and 12 weeks (week 18) post-intervention.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 42
Watts
  Workstream 1 - baseline peak power output: number analyzed (Participants) | 13
  Workstream 1 - baseline peak power output | 94.9 (26.1)
  Workstream - 1 post-intervention peak power output: number analyzed (Participants) | 13
  Workstream - 1 post-intervention peak power output | 103.7 (30.4)
  Workstream 1 - 4-weeks post-intervention follow-up peak power output: number analyzed (Participants) | 10
  Workstream 1 - 4-weeks post-intervention follow-up peak power output | 98.7 (23.4)
  Workstream 1 - 12-week post-intervention follow-up peak power output: number analyzed (Participants) | 9
  Workstream 1 - 12-week post-intervention follow-up peak power output | 102.7 (30.8)
  Workstream 2 - baseline peak power output: number analyzed (Participants) | 29
  Workstream 2 - baseline peak power output | 101.6 (39.4)
  Workstream 2 - post-intervention follow-up peak power output: number analyzed (Participants) | 29
  Workstream 2 - post-intervention follow-up peak power output | 106.0 (43.0)
  Workstream 2 - 4-weeks post-intervention follow-up peak power output: number analyzed (Participants) | 16
  Workstream 2 - 4-weeks post-intervention follow-up peak power output | 112.0 (44.5)
  Workstream 2 - 12-weeks post-intervention follow-up peak power output: number analyzed (Participants) | 20
  Workstream 2 - 12-weeks post-intervention follow-up peak power output | 114.1 (45.5)

14. Secondary Outcome: Pain-free Walking Distance
Description: assessment of the distance that the patient can currently walk before experiencing claudication pain.
Time Frame: Baseline, post-intervention (week 6), then 4 weeks (week 10) and 12 weeks (week 18) post-intervention.
Population: Only patients completing the programme and providing baseline and follow-up data are included. This comprises:
  Post-intervention follow-up Workstream 1; n = 15/30 Workstream 2; n = 30/40 Total = 45/70.
  4-week post-intervention follow-up Workstream 1; n = 12/30 Workstream 2; n = 16/40 Total = 28/70.
  12-week post-intervention follow-up Workstream 1; n =11/30 Workstream 2; n = 24/40 Total = 35/70.
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 45
metres
  Workstream 1 baseline: number analyzed (Participants) | 15
  Workstream 1 baseline | 114.1 (75.4)
  Workstream 1 Post-intervention follow-up: number analyzed (Participants) | 15
  Workstream 1 Post-intervention follow-up | 141.3 (62.4)
  Workstream 1 - 4-week post intervention follow-up: number analyzed (Participants) | 12
  Workstream 1 - 4-week post intervention follow-up | 172.4 (103.5)
  Workstream 1 - 12-week post intervention follow-up: number analyzed (Participants) | 11
  Workstream 1 - 12-week post intervention follow-up | 216.3 (163.2)
  Workstream 2 baseline: number analyzed (Participants) | 30
  Workstream 2 baseline | 142.5 (95.5)
  Workstream 2 Post-intervention follow-up: number analyzed (Participants) | 30
  Workstream 2 Post-intervention follow-up | 218.6 (166.6)
  Workstream 2 - 4-week post intervention follow-up: number analyzed (Participants) | 16
  Workstream 2 - 4-week post intervention follow-up | 212.7 (173.8)
  Workstream 2 - 12-week post intervention follow-up: number analyzed (Participants) | 24
  Workstream 2 - 12-week post intervention follow-up | 276.0 (214.7)

15. Secondary Outcome: Ventilatory Anaerobic Threshold (VAT)
Description: Ventilatory anaerobic threshold assessed via cardiopulmonary exercise testing
Time Frame: Baseline, post-intervention (week 6), then 4 weeks (week 10) and 12 weeks (week 18) post-intervention.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 42
ml/kg/min
  Workstream 1 - baseline VAT: number analyzed (Participants) | 13
  Workstream 1 - baseline VAT | 9.8 (1.7)
  Workstream 1 - post-intervention follow-up VAT: number analyzed (Participants) | 13
  Workstream 1 - post-intervention follow-up VAT | 10.2 (1.7)
  Workstream 1 - 4-week post-intervention follow-up VAT: number analyzed (Participants) | 10
  Workstream 1 - 4-week post-intervention follow-up VAT | 10.0 (1.3)
  Workstream 1 - 12-week post-intervention follow-up VAT: number analyzed (Participants) | 9
  Workstream 1 - 12-week post-intervention follow-up VAT | 9.4 (1.4)
  Workstream 2 - baseline VAT: number analyzed (Participants) | 29
  Workstream 2 - baseline VAT | 10.0 (1.9)
  Workstream 2 - post-intervention follow-up VAT: number analyzed (Participants) | 29
  Workstream 2 - post-intervention follow-up VAT | 10.4 (2.2)
  Workstream 2 - 4-week post-intervention follow-up VAT: number analyzed (Participants) | 16
  Workstream 2 - 4-week post-intervention follow-up VAT | 9.8 (2.1)
  Workstream 2 - 12-week post-intervention follow-up VAT: number analyzed (Participants) | 20
  Workstream 2 - 12-week post-intervention follow-up VAT | 10.1 (2.2)

16. Secondary Outcome: Quality of Life Questionnaire Short-form-36 (SF-36)
Description: as for outcome 10
Time Frame: 4 weeks (week 10) and 12 weeks (week 18) post-intervention
Population: Only patients completing the programme and providing baseline and follow-up data are included. This comprises:
  4-week follow-up: Workstream 1; n = 13/30 Workstream 2; n = 16/40 Total = 29/70.
  12-week follow-up: Workstream 1; n = 11/30 Workstream 2; n = 24/40 Total = 35/70.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 35
units on a scale
  Workstream 1 - 4-week follow-up physical functioning: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up physical functioning | 61.9 (20.1)
  Workstream 1 - 12-week follow-up physical functioning: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up physical functioning | 64.1 (20.2)
  Workstream 1 - 4-week follow-up role physical: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up role physical | 61.5 (30.9)
  Workstream 1 - 12-week follow-up follow-up role physical: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up follow-up role physical | 62.5 (26.8)
  Workstream 1 - 4-week follow-up pain: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up pain | 53.2 (19.6)
  Workstream 1 - 12-week follow-up pain: number analyzed (Participants) | 10
  Workstream 1 - 12-week follow-up pain | 54.1 (24.7)
  Workstream 1 - 4-week follow-up general health: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up general health | 47.4 (13.9)
  Workstream 1 - 12-week follow-up general health: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up general health | 53.5 (19.3)
  Workstream 1 - 4-week follow-up vitality: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up vitality | 51.0 (17.5)
  Workstream 1 - 12-week follow-up vitality: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up vitality | 55.1 (7.3)
  Workstream 1 - 4-week follow-up social functioning: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up social functioning | 84.6 (20.5)
  Workstream 1 - 12-week follow-up social functioning: number analyzed (Participants) | 10
  Workstream 1 - 12-week follow-up social functioning | 85.0 (17.5)
  Workstream 1 - 4-week follow-up role emotional: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up role emotional | 80.8 (31.6)
  Workstream 1 - 12-week follow-up role emotional: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up role emotional | 76.5 (23.8)
  Workstream 1 - 4-week follow-up mental health: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up mental health | 71.2 (15.2)
  Workstream 1 - 12-week follow-up mental health: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up mental health | 71.8 (15.2)
  Workstream 1 - 4-week follow-up PCS: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up PCS | 40.9 (8.4)
  Workstream 1 - 12-week follow-up PCS: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up PCS | 38.8 (15.4)
  Workstream 1 - 4 week follow-up MCS: number analyzed (Participants) | 13
  Workstream 1 - 4 week follow-up MCS | 51.5 (9.3)
  Workstream 1 - 12-week follow-up MCS: number analyzed (Participants) | 11
  Workstream 1 - 12-week follow-up MCS | 46.8 (17.3)
  Workstream 2 - 4-week follow-up physical functioning: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up physical functioning | 61.7 (19.9)
  Workstream 2 - 12-week follow-up physical functioning: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up physical functioning | 61.5 (20.3)
  Workstream 2 - 4-week follow-up role physical: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up role physical | 63.9 (24.5)
  Workstream 2 - 12-week follow-up role physical: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up role physical | 57.3 (23.4)
  Workstream 2 - 4-week pain: number analyzed (Participants) | 16
  Workstream 2 - 4-week pain | 55.6 (20.3)
  Workstream 2 - 12-week follow-up pain: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up pain | 57.5 (23.6)
  Workstream 2 - 4-week follow-up general health: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up general health | 54.6 (18.1)
  Workstream 2 - 12-week follow-up general health: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up general health | 53.2 (19.5)
  Workstream 2 - 4-week follow-up vitality: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up vitality | 54.9 (20.7)
  Workstream 2 - 12 -week follow-up vitality: number analyzed (Participants) | 24
  Workstream 2 - 12 -week follow-up vitality | 54.8 (22.0)
  Workstream 2 - 4-week follow-up social functioning: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up social functioning | 79.9 (25.4)
  Workstream 2 - 12-week follow-up social functioning: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up social functioning | 76.5 (27.8)
  Workstream 2 4-week follow-up role emotional: number analyzed (Participants) | 16
  Workstream 2 4-week follow-up role emotional | 77.3 (26.5)
  Workstream 2 - 12-week follow-up role emotional: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up role emotional | 77.7 (26.5)
  Workstream 2 4-week follow-up mental health: number analyzed (Participants) | 16
  Workstream 2 4-week follow-up mental health | 78.9 (17.4)
  Workstream 2 - 12-week follow-up mental health: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up mental health | 78.0 (18.6)
  Workstream 2 - 4-week follow-up PCS: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up PCS | 41.7 (7.5)
  Workstream 2 - 12-week follow-up PCS: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up PCS | 41.0 (8.6)
  Workstream 2 - 4-week follow-up MCS: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up MCS | 52.5 (10.0)
  Workstream 2 - 12-week follow-up MCS: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up MCS | 52.3 (11.2)

17. Secondary Outcome: Vascular Quality of Life Questionnaire - (VascuQol)
Description: as for outcome 11
Time Frame: 4 weeks (week 10) and 12 weeks (week 18) post-intervention.
Population: Only patients completing the programme and providing follow-up data are included. This comprises:
  4-week follow-up: Workstream 1; n = 13/30 Workstream 2; n = 16/40 Total = 29/70. 12-week follow-up: Workstream 1; n = 10/30 Workstream 2; n = 24/40 Total = 34/70.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High-Intensity Interval Training
Number analyzed (Participants) | 34
units on a scale
  Workstream 1 - 4-week follow-up pain score: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up pain score | 4.7 (1.7)
  Workstream 1 -12-week follow-up pain score: number analyzed (Participants) | 10
  Workstream 1 -12-week follow-up pain score | 5.4 (1.2)
  Workstream 1 - 4-week follow-up social score: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up social score | 6.3 (1.1)
  Workstream 1 - 12-week follow-up social score: number analyzed (Participants) | 10
  Workstream 1 - 12-week follow-up social score | 6.4 (0.9)
  Workstream 1 - 4-week follow-up activities score: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up activities score | 5.2 (1.0)
  Workstream 1 - 12-week follow-up activities score: number analyzed (Participants) | 10
  Workstream 1 - 12-week follow-up activities score | 5.2 (1.2)
  Workstream 1 - 4-week follow-up symptom score: number analyzed (Participants) | 13
  Workstream 1 - 4-week follow-up symptom score | 5.8 (0.6)
  Workstream 1 - 12-week follow-up symptom score: number analyzed (Participants) | 10
  Workstream 1 - 12-week follow-up symptom score | 5.9 (0.7)
  Workstream 1 4-week follow-up emotional score: number analyzed (Participants) | 13
  Workstream 1 4-week follow-up emotional score | 6.0 (1.0)
  Workstream 1 - 12-week follow-up emotional score: number analyzed (Participants) | 10
  Workstream 1 - 12-week follow-up emotional score | 6.4 (0.4)
  Workstream 1 - 4-week total score: number analyzed (Participants) | 13
  Workstream 1 - 4-week total score | 5.6 (1.0)
  Workstream 1 - 12-week follow-up total score: number analyzed (Participants) | 10
  Workstream 1 - 12-week follow-up total score | 5.8 (0.7)
  Workstream 2 4-week follow-up pain score: number analyzed (Participants) | 16
  Workstream 2 4-week follow-up pain score | 4.8 (1.3)
  Workstream 2 - 12-week follow-up pain score: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up pain score | 4.6 (1.3)
  Workstream 2 - 4-week follow-up social score: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up social score | 5.5 (1.6)
  Workstream 2 - 12-week follow-up social score: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up social score | 5.4 (1.7)
  Workstream 2 4-week follow-up activities score: number analyzed (Participants) | 16
  Workstream 2 4-week follow-up activities score | 4.9 (1.2)
  Workstream 2 - 12-week follow-up activities score: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up activities score | 4.7 (1.1)
  Workstream 2 4-week follow-up symptom score: number analyzed (Participants) | 16
  Workstream 2 4-week follow-up symptom score | 5.3 (1.2)
  Workstream 2 - 12-week follow-up symptom score: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up symptom score | 5.2 (1.2)
  Workstream 2 4-week follow-up emotional score: number analyzed (Participants) | 16
  Workstream 2 4-week follow-up emotional score | 5.7 (1.3)
  Workstream 2 - 12-week follow-up emotional score: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up emotional score | 5.5 (1.1)
  Workstream 2 - 4-week follow-up total score: number analyzed (Participants) | 16
  Workstream 2 - 4-week follow-up total score | 5.2 (1.2)
  Workstream 2 - 12-week follow-up total score: number analyzed (Participants) | 24
  Workstream 2 - 12-week follow-up total score | 5.0 (1.1)

ADVERSE EVENTS:
Time Frame: From enrollment to 18 weeks later for each patient.
Arm/Group | High-Intensity Interval Training
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 1/70
Other Adverse Events (participants affected / at risk) | 10/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Intensity Interval Training (N=70)
Thrombosed popliteal aneurysm (Vascular disorders) | 1 (1) — The SAE was a thrombosed popliteal aneurysm that occurred in the period between two exercise sessions. The patient was admitted for surgery and underwent a lower limb bypass procedure. Symptoms occurred 2 days after exercise so unlikely related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Intensity Interval Training (N=70)
Post-exercise dizzines (General disorders) | 6 (7) — There were 7 occurrences of dizziness that occurred after exercise sessions or CPET
Dull chest ache (Cardiac disorders) | 1 (1) — an isolated episode of a 'dull chest ache' that occurred in the period between two exercise sessions. Following referral to cardiology a diagnosis of probable angina was made but not confirmed as a diagnostic angiogram was refused.
Back spasm (Musculoskeletal and connective tissue disorders) | 1 (1) — The occurrence of a back spasm after an exercise session.
Headache (General disorders) | 1 (1) — One occurrence of a headache after exercise
Hypertensive CPET response (Cardiac disorders) | 1 (1) — One occurrence of a hypertensive CPET response

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT04042311/Prot_SAP_000.pdf